CLINICAL TRIAL: NCT05111665
Title: The Association Between Decentering and Reductions in Relapse/Recurrence in Mindfulness-Based Cognitive Therapy for Depression in Adults: A Randomized Controlled Trial
Brief Title: Decentering and Relapse/Recurrence in MBCT for Depression in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Mark Lau, Principle Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H07-03046
Record Dates: First submitted 2021-10-04; First posted 2021-11-08 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: Depression; Depressive Disorder, Major; Depression in Remission
MeSH Terms: conditions — Depression; Depressive Disorder, Major | interventions — Mindfulness-Based Cognitive Therapy; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mindfulness-based Cognitive Therapy (MBCT) (Experimental): Remitted depressed participants received eight-weekly, two-hour MBCT sessions (Segal et al., 2013). This program combines MBSR meditation practices (e.g., body scan, mindful stretching, mindfulness of breath/body/sounds/thoughts) with traditional CT techniques (e.g., psychoeducation about depression symptoms and automatic thoughts, exercises designed to demonstrate how the nature of one's thoughts change with one's mood, questioning of automatic thoughts and creating a relapse prevention plan). Finally, participants engaged in a daily meditation practice and homework exercises directed at integrating the application of awareness skills into daily life. Each MBCT group was led by a masters-level clinician who was an active MBCT/Mindfulness-Based Stress Reduction (MBSR) instructor.
  Interventions: Behavioral: Mindfulness-based Cognitive Therapy (MBCT)
- Relaxation Group Therapy (RGT) (Active Comparator): The revised edition of the Changeways Relaxation Programme (Paterson, 1997) served as the active control condition to control for non-specific group factors including group participation, expectation of change or therapeutic contact and attention. The rationale was that relaxation can be used to better manage life stressors which precipitate depressive episodes. Participants received eight-weekly, two-hour relaxation training sessions. This group program combines psychoeducation regarding the effects of stress, diaphragmatic breathing, progressive muscle relaxation, passive relaxation and imagery. It also incorporates time for participants to discuss the events of the week to facilitate the supportive aspect of group participation. Finally, participants were asked to engage in daily exercises to practice the various relaxation strategies. Each RGT group was led by a doctoral-level therapist.
  Interventions: Behavioral: Relaxation Group Therapy (RGT)
- Treatment as usual (TAU) (Placebo Comparator): Participants randomized to the TAU group were instructed that participants would receive MBCT at the end of the follow-up period and to seek help from their family doctors or other sources as the normally would, should the participants encounter symptomatic deterioration or other difficulties over the course of the study. At the end of the follow-up phase, participants in the TAU and RGT group were offered the opportunity to receive MBCT.
  Interventions: Behavioral: Treatment as usual (TAU)

INTERVENTIONS:
Behavioral: Mindfulness-based Cognitive Therapy (MBCT)
  Arms: Mindfulness-based Cognitive Therapy (MBCT)
Behavioral: Relaxation Group Therapy (RGT)
  Arms: Relaxation Group Therapy (RGT)
Behavioral: Treatment as usual (TAU)
  Arms: Treatment as usual (TAU)

SUMMARY:
Objective: "Decentering" is defined as the ability to observe one's thoughts and feelings as temporary, objective events in the mind, and is increasingly regarded as a candidate mechanism in mindfulness-based interventions. The current study sought to examine the role of decentering, and other related variables, in the efficacy of Mindfulness-based cognitive therapy (MBCT) as compared to two active comparison conditions.

Method: Formerly depressed individuals (N = 227), randomly assigned to MBCT (n = 74), relaxation group therapy (RGT; n = 77) or treatment-as-usual (TAU; n = 76), completed self-report measures of decentering and symptoms of depression at pre-, mid-, and post-treatment, and relapse was assessed at 3, 6, 9, and 12 months, post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* a Diagnostic and Statistical Manual of Mental Disorders (4th ed.; DSM IV-TR; American Psychiatric Association (APA), diagnosis of major depressive disorder (MDD) without psychotic features, in Full Remission;
* three or more prior major depressive episodes;
* age between 18 and 65 years;
* cognitive reactivity (CR) or mood-activated dysfunctional beliefs score greater than or equal to eight (see assessment procedure below);
* a score of less than 10 on the Hamilton Rating Scale for Depression (HRSD);
* minimum of a 10 week period free of psychotropic medication other than stable dosage of antidepressant medication for a minimum of four weeks;
* fluency in English; An increased cognitive reactivity score of eight points or more and,
* ability to give informed consent and complete questionnaires unassisted.

Exclusion Criteria:

* a diagnosis of bipolar disorder (past or present), schizophreniform disorders, substance abuse or dependence (current or within the past six months), borderline or antisocial personality disorder, or neurocognitive disorders;
* current psychotherapy or counselling more frequently than twice per month;
* current practice of meditation more than once per week or yoga more than twice per week;
* electroconvulsive therapy within the past six months; or
* self-reported ingestion of alcohol or other psychoactive substances within the past 48 hrs.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2008-02-14 (Actual); Primary Completion 2008-10-31 (Actual); Study Completion 2008-10-31 (Actual)

PRIMARY OUTCOMES:
Major depressive disorder (MDD) relapse/recurrence - incidence of | 12- month post-treatment follow-up
  Number of participants meeting criteria for relapse/recurrence of MDD during follow-up
Change in major depressive disorder (MDD) relapse/recurrence - time to relapse/recurrence | 3-, 6-, 9-, and 12- month post-treatment follow-up
  Change in relapse/recurrence of MDD (i.e., survival) across follow-up

SECONDARY OUTCOMES:
Change in Beck Depression Inventory - Second Edition total scores | Pre-, mid- (i.e., at week 4 of MBCT), and post-treatment (i.e., after 8 weeks of MBCT)
  Change in symptoms of depression across MBCT treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Mark Lau, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Moore MT, Lau MA, Haigh EAP, Willett BR, Bosma CM, Fresco DM. Association between decentering and reductions in relapse/recurrence in mindfulness-based cognitive therapy for depression in adults: A randomized controlled trial. J Consult Clin Psychol. 2022 Feb;90(2):137-147. doi: 10.1037/ccp0000718. PMID 35343725